CLINICAL TRIAL: NCT06284005
Title: Multicentre Interventional Pilot Study on the Evaluation of the Functionality, Safety and Reliability of a New Robotic Prosthesis for the Lower Limb At the Transfemoral Level
Brief Title: Study on the Functionality, Safety and Reliability of a Robotic Prosthesis for the Lower Limb At the Transfemoral Level
Acronym: MOTU-ATP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Claudio Macchi, Full Professor, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MOTU ATP - Studio clinico
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Amputation; Traumatic Amputation; Leg Injury; Lower Limb Injury
Keywords: lower limb; transfemoral
MeSH Terms: conditions — Amputation, Traumatic; Leg Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prosthetic group (Experimental): prosthetic group performs the entire protocol with the prosthesis prototype.
  Interventions: Device: WRL ATP

INTERVENTIONS:
Device: WRL ATP — evaluation of functionality, degree of safety and reliability of the lower limb prosthesis prototype

SUMMARY:
The goal of this multicenter interventional pilot is to verify the functionality of a prosthesis for trans-femoral amputees.

The main question it aims to answer are:

* Is to verify the technical functionality, safety and reliability of the propulsive lower limb prosthesis prototype, with active ankle, so as to provide indications regarding the technical and functional developments to be implemented in the finalization of the device.
* Provide an indication of the functional effectiveness of the device and its satisfaction by patients.

Participants will perform:

* walking tests inside parallel bars on flat and/or inclined terrain;
* walking tests on treadmill;
* stair climbing/descent tests.

ELIGIBILITY:
Inclusion Criteria:

* trans femoural amputation
* Medicare Functional Classification Levels k3-k4
* expert prosthesis wearer (more than one year)
* electronic knee prostheses user
* energy-release prosthetic foot user

Exclusion Criteria:

* Relevant medical comorbidities
* heart device wearers (PMK or AICD)
* cognitive impairment
* anxious or depressed illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
ad hoc check-list Adverse Event | baseline
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 2
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 3
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 4
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
ad hoc check-list Adverse Event | day 5
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: claudio macchi, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gailey R, Allen K, Castles J, Kucharik J, Roeder M. Review of secondary physical conditions associated with lower-limb amputation and long-term prosthesis use. J Rehabil Res Dev. 2008;45(1):15-29. doi: 10.1682/jrrd.2006.11.0147. PMID 18566923
- [Background] Mak AF, Zhang M, Boone DA. State-of-the-art research in lower-limb prosthetic biomechanics-socket interface: a review. J Rehabil Res Dev. 2001 Mar-Apr;38(2):161-74. PMID 11392649
- [Background] Pirouzi G, Abu Osman NA, Eshraghi A, Ali S, Gholizadeh H, Wan Abas WA. Review of the socket design and interface pressure measurement for transtibial prosthesis. ScientificWorldJournal. 2014;2014:849073. doi: 10.1155/2014/849073. Epub 2014 Aug 13. PMID 25197716
- [Background] Segal AD, Orendurff MS, Klute GK, McDowell ML, Pecoraro JA, Shofer J, Czerniecki JM. Kinematic and kinetic comparisons of transfemoral amputee gait using C-Leg and Mauch SNS prosthetic knees. J Rehabil Res Dev. 2006 Nov-Dec;43(7):857-70. doi: 10.1682/jrrd.2005.09.0147. PMID 17436172